CLINICAL TRIAL: NCT06378320
Title: eHealth for Breastfeeding Support - the HOTSPOT Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Lydia Furman, Attending Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20240287
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Feeding
Keywords: African American; Smartphone app; Milk, Human
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This will be a prospective randomized two arm study for expectant women and a prospective randomized two arm study for fathers/partners. All participants receive access to the wireframe app. Maternal participants will be randomized to nudge or no nudge via text with those in the app "nudge" group receiving questions weekly prior to delivery and biweekly (every 2 weeks) after delivery through 3 months postpartum. The purpose of these "nudges" is to assess whether participants are more likely to access and benefit from the app if they are encouraged to explore it. Father/partner participants will also be randomized to either a nudge or no nudge group with those in the "nudge" group receiving questions weekly for the first two months and then biweekly (every 2 weeks) for another two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Maternal participants nudge group (Experimental): Participants in the app "nudge" group receive access to the app and questions with app cues by text weekly prior to delivery and biweekly (every 2 weeks) after delivery through 3 months postpartum.
  Interventions: Other: App access and Text message
- Maternal participants no nudge group (Other): Participants in the app "no nudge" group receive access to the app and no questions with app cues through 3 months postpartum.
  Interventions: Other: App access only
- Father/partner participants nudge group (Experimental): Participants in the app "nudge" group receive access to the app and questions with app cues by text weekly for the first 2 months and then biweekly (every 2 weeks) for another 2 months.
  Interventions: Other: App access and Text message
- Father/partner participants no nudge group (Other): Participants in the app "no nudge" group receive access to the app and no questions with app cues for 4 months.
  Interventions: Other: App access only

INTERVENTIONS:
Other: App access and Text message — Access to App and Text messages with app related breastfeeding related question
  Other Names: App access and Text nudge
  Arms: Father/partner participants nudge group; Maternal participants nudge group
Other: App access only — Access to App without Text messages with app related breastfeeding related question
  Other Names: App access
  Arms: Father/partner participants no nudge group; Maternal participants no nudge group

SUMMARY:
This is a voluntary research study to test use of a phone app that is intended to support breastfeeding specifically for African American and Black people. This is called a "pilot" study because the app is still in development. The goal of this research is to see if mothers use the app more when they receive text "nudges" to look at it compared to not getting those "nudges". The research project is being conducted by Lydia Furman MD.

The purpose of the app (which is currently in clickable "wireframe" status, a "pre" app phase) is to support and promote breastfeeding specifically for mothers and fathers/partners who are African American or Black. Other breastfeeding apps have pictures mainly of White or Asian mothers and information that is not oriented toward African American mothers. This app aims to provide accurate and needed breastfeeding information that is culturally attuned.

Up to 24 participants will be enrolled at UHCMC, including up to 20 mothers. Other participants will include up to 4 African American or Black fathers/partners whose partners are interested in breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Maternal participants
* Adult women who are expecting (pregnant) and between 24-34 weeks gestation
* Self-describe as African-American or Black (AA/B)
* Have a smart phone
* Receive prenatal care at either Ahuja Rainbow Center for Women and Children or MacDonald and Women's Suite 1200 at University Hospitals
* Either interested in or committed to breastfeeding for their infant
* Father/partner participants
* Father (mother/partner is expectant or delivered) or plan to become father
* Age 18 years or older
* Have a smart phone or a personal device or iPad
* Attending programming at Passages, Inc.
* Self-identified interest in how their own infant will be fed
* Self-describe as African-American or Black

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Potential participants may enroll as expectant women or as a father/partner. Gender is self-identified.
Enrollment: 20 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Maternal participants app usability score | Up to 3 months postpartum
  Percentage of participants with System Usability Scale score of >78.8
Father/partner participants app usability score | Up to 4 months post-enrollment
  Percentage of participants with System Usability Scale score of >78.8
Maternal participants app engagement score | Up to 3 months postpartum
  Percentage of participants with an app interaction score of more than 1 on a 5 point scale with 1 meaning no engagement past week and 5 meaning more than daily engagement in the past week
Father/partner participants app engagement score | Up to 4 months post-enrollment
  Percentage of participants with an app interaction score of more than 1 on a 5 point scale with 1 meaning no engagement past week and 5 meaning more than daily engagement in the past week

SECONDARY OUTCOMES:
Maternal participants breastfeeding knowledge at enrollment | At enrollment
  Percentage of participants with 75% or more correct responses to 4 breastfeeding knowledge questions
Maternal participants breastfeeding knowledge after app exposure | At 2 months postpartum
  Percentage of participants with 75% or more correct responses to 10 breastfeeding
Father/partner participants breastfeeding knowledge at enrollment | At enrollment
  Percentage of participants with 75% or more correct responses to 4 breastfeeding knowledge questions
Father/partner participants breastfeeding knowledge after app exposure | At 3 months post-enrollment
  Percentage of participants with 75% or more correct responses to 10 breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Furman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (3):
- United States (3):
  - Ahuja Rainbow Center for Women and Children, Cleveland, Ohio
  - Passages, Inc., Cleveland, Ohio
  - University Hospital MacDonald Women's Hospital, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No